CLINICAL TRIAL: NCT05276947
Title: The Effect of Peanut Ball Use on Labor Process and Maternal - Neonatal Outcomes in Obese Pregnants
Brief Title: The Use of Peanut Ball in Labor in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Fulden Ozkececi, Principal Investigator, Gulhane Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PBinON
Record Dates: First submitted 2022-02-07; First posted 2022-03-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Labor Long
Keywords: Peanut ball
MeSH Terms: interventions — Patient Positioning

STUDY DESIGN:
Intervention Model Description: There will be an intervention group and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peanut ball intervention (Experimental): The experimental group. In the active phase of the labor (cervical dilatation = 5 cm), the peanut ball, which has a cover provided by the researcher and changed in each patient, will be placed between the knees of the participant for at least 30 minutes every hour, and a position change will be provided with the peanut ball in each time. The positions to be given with the peanut ball, semi sitting lunge, side lying, tucked, leaning forward, pushing and sitting position.
  Interventions: Other: position with peanut ball
- Control group (No Intervention): Standard care will be given to the control group without positioning with a peanut ball.

INTERVENTIONS:
Other: position with peanut ball — The experimental group will be positioned with the peanut ball until the end of the active phase of labor.
  Arms: Peanut ball intervention

SUMMARY:
The purpose of this study is to assess the efficacy of peanut ball use on labor process and maternal, neonatal outcomes in obese pregnant women.

DETAILED DESCRIPTION:
After being informed about the study, all participants giving written informed consent, on the active phase of labor (cervical dilatation = 5 cm), the pregnant women in the experimental group will be provided with a position change lasting at least 30 minutes every hour with a peanut ball. The peanut ball will be used with a sheath that is changed for each participant. Pregnant women in the control group will be included in the study during the active phase of labor (cervical dilatation = 5 cm). No intervention will be made by the researcher. They will receive standard care by the service nurse.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for delivery
* Maternal BMI > 30kg/m2 at admission
* Gestational age > 37 weeks 0 days
* Singleton pregnancy
* Cephalic presentation
* Cervical dilatation less than 5 cm
* Turkish speaking

Exclusion Criteria:

* Pre-pregnancy BMI < 30kg/m2
* Gestational age < 37 weeks 0 days
* Multifetal gestation
* Intrauterine fetal demise
* Musculoskeletal problems
* Receiving magnesium sulfate
* High risk pregnancies (Preeclampsia/eclampsia, cholestasis, intrauterine growth retardation, fetal anomaly, polyhydramnios or oligohydramnios)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-08-13 (Actual); Study Completion 2023-08-13 (Actual)

PRIMARY OUTCOMES:
Labor time | From 5 cm of cervical dilatation to the second stage of labor
  The primary outcome measure is the length of first stage (active phase) and second stage of labor in obese pregnant women.

SECONDARY OUTCOMES:
Pain level | Latent phase, active phase and at cervical dilatation 10 cm (on contractions)
  Visual Analog Scale (VAS) is used to convert some values that cannot be measured numerically. Two end definitions of the parameter to be evaluated are written at the two ends of a 10 cm line, and the patient is asked to indicate where on this line their situation is appropriate by drawing a line or by placing a dot or pointing. For example, for pain, I have no pain at one end and very severe pain at the other end and the patient marks his/her current state on this line. The length of the distance from the point where there is no pain to the point marked by the patient indicates the patient's pain (0: no pain 10: severe pain)
Operative vaginal delivery rate | From 5 cm of cervical dilatation to the expulsion phase of labor
  Forceps/vacuum
Type of delivery | From 5 cm of cervical dilatation to the expulsion phase of labor
  Cesarean section or vaginal delivery
Maternal complications | From 5 cm of cervical dilatation to the expulsion phase of labor
  Perineal laceration and atony
Neonatal complications | From 5 cm of cervical dilatation to the expulsion phase of labor
  APGAR score, need for neonatal intensive care. For the Apgar score, five symptoms are checked, including respiration, heart rate, color, tone, and response to stimuli. Each symptom is scored as 0, 1, or 2. The baby is scored as '0' if there is no breathing or heartbeat, his color is pale or cyanotic, his tone is loose, and he does not respond to the stimulus given by inserting the catheter into the nose.
Birth satisfaction | Postpartum first hour
  Birth Satisfaction Scale A minimum of 30 and a maximum of 150 points are obtained from the scale. The higher the score, the higher the level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Gulten GUVENC, PhD, RN, Study Director — Gulhane Faculty of Nursing, University of Health Sciences
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No